CLINICAL TRIAL: NCT06641596
Title: Effects of Chromium, Phyllanthus Emblica Fruit Extract, and Shilajit Supplementation on Markers of Cardiovascular Health, Fitness, and Weight Loss in Men and Women Initiating an Exercise and Diet Intervention Program
Brief Title: Impact of Chromium, Phyllanthus Emblica, and Shilajit on Cardiovascular Health, Fitness, and Weight Loss During Exercise and Diet Programs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kerry Group P.L.C (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: S23-1467336
Record Dates: First submitted 2024-09-11; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Overweight; Metabolic Syndrome X
MeSH Terms: conditions — Overweight; Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: 24 participants per group equally comprised of men and women matched as closely as possible by age, gender, BMI, and body mass
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Placebo (Placebo Comparator): 2 x 500 mg capsules
  Interventions: Dietary Supplement: Placebo
- Dietary Supplement 1 (Experimental): 1 x 20 mg capsule of Cr-400 (formulation of 400 mcg of trivalent chromium with 6 mg of PE and 6 mg of SJ) + 1x500 capsule of PLA
  Interventions: Dietary Supplement: Cr-400
- Dietary Supplement 2 (Experimental): 2 x 20 mg capsule of Cr-400 (formulation of 400 mcg of trivalent chromium with 6 mg of PE and 6 mg of SJ)
  Interventions: Dietary Supplement: Cr-800
- Dietary Supplement 3 (Experimental): 1 x 500 mg capsule of PE (500mg) + 1 x 500 mg capsule of PLA
  Interventions: Dietary Supplement: PE-500
- Dietary Supplement 4 (Experimental): 2 x 500 mg capsules of PE (1000 mg)
  Interventions: Dietary Supplement: PE-1000

INTERVENTIONS:
Dietary Supplement: Placebo — 2 capsules of Placebo, once daily after breakfast for 12 weeks
  Arms: Placebo
Dietary Supplement: Cr-400 — 1 capsule of Cr-400 + 1 capsule of Placebo, once a day after breakfast for 12 weeks
  Arms: Dietary Supplement 1
Dietary Supplement: Cr-800 — 2 capsules of Cr-400, once a day after breakfast for 12 weeks
  Arms: Dietary Supplement 2
Dietary Supplement: PE-500 — 1 capsule of PE + 1 capsule of Placebo, once a day after breakfast for 12 weeks
  Arms: Dietary Supplement 3
Dietary Supplement: PE-1000 — 2 capsules of PE-500, once a day after breakfast for 12 weeks
  Arms: Dietary Supplement 4

SUMMARY:
A randomized, double-blind, placebo controlled, parallel study to determine if Chromium (Cr), Phyllanthus emblica (PE) and Shilajit (SJ) supplementation and Phyllanthus emblica fruit extract supplementation promotes greater changes in glucose homeostasis, endothelial function, and cardiometabolic risk in sedentary and overweight men and women initiating an exercise and weight loss program.

DETAILED DESCRIPTION:
Men and women with at least 2 markers of metabolic syndrome will participate in a randomized, placebo-controlled, parallel, and repeated measures intervention trial. Volunteers will participate in a standardized resistance training (3 sessions/week) and aerobic training (3 x 30 min sessions/week) program while reducing energy intake by 5 kcals/kg/d.

In a double-blind and randomized manner, participants will be matched by age, sex, BMI, and body mass to supplement their diet with placebo (PLA), 400 mcg of trivalent chromium with 6 mg of PE and 6 mg of SJ (Cr-400), or 800 mcg of trivalent chromium with 12 mg of PE and 12 mg of SJ (Cr-800), or 500 mg of PE (PE-500), or 1000 mg of PE (PE-1000) once a day after breakfast for 12-weeks.

Fasting blood samples, DEXA body composition, platelet aggregation, and ultrasound flow-mediated dilation (FMD) studies will be conducted at 0, 6, and 12 weeks of supplementation.

ELIGIBILITY:
Inclusion Criteria:

1. Sedentary males and females age 30-65 years with a BMI >30 and/or percent body fat >30%
2. Medical clearance for participating in moderate to intense exercise training and testing;
3. meet the 2006 International Diabetes Federation criteria for central obesity (ethnicity specific waist circumference) and any two risk factors to metabolic syndrome (i.e., fasting triglycerides > 150 mg/dL or treatment for high triglycerides, HDL <40 mg/dL in males and <50 mg/dL in female, resting SBP >130 mmHg or DBP >85 mmHg or treatment of previously diagnosed hypertension, blood glucose ≥ 100 mg/dl or previous diagnosis for Type II diabetes);
4. Absence of limiting musculoskeletal injury that would prevent participation in a general fitness program; and,
5. Has given voluntary, written, informed consent to participate in the study.

Exclusion Criteria:

Participants will not be allowed to participate in the study if:

1. they currently take or have taken nitrous oxide or anti-inflammatory type supplements or medications within one month of the start of the study;
2. they have uncontrolled hypertension, triglycerides >500 mg/dL, elevated AST and ALT > 3 times the upper limit, and serum creatinine >1.5 mg/dL);
3. They do not receive medical clearance from their personal physician to participate in the study and exercise program;
4. They are pregnant or plan to become pregnant; and/or
5. They are unable to complete at least 90% of the training.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-05-29 (Actual)

PRIMARY OUTCOMES:
Flow-Mediated Dilation (FMD) | Baseline, 6 and 12 weeks
  Percentage of change in the Flow-Mediated Dilation (FMD).
Venous Occlusion (VO) | Baseline, 6 and 12 weeks
  Changes in the Venous Occlusion (VO) for the FMD cuff: mmHg
Platelet Aggregation | Baseline, 6 and 12 weeks
  Check participants' Platelet Aggregation (Ohms)
Fasting Glucose | Baseline, 6 and 12 weeks
  To assess changes in participants' levels of fasting glucose (mg/dL)
HbA1c | Baseline, 6 and 12 weeks
  To assess changes in the concentration of HbA1c (mmol/mol)
C-reactive protein (CRP) | Baseline, 6 and 12 weeks
  To assess changes in the level of CRP (mg/L)
Lipid Profile-Cholesterol | Baseline, 6 weeks and 12 weeks
  Changes in the level of cholesterol (mg/dL)
Lipid Profile -Triglycerides | Baseline, 6 weeks and 12 weeks
  Changes in the level of Triglycerides (mg/dL)
Lipid Profile- HDL Cholesterol | Baseline, 6 and 12 weeks
  Changes in the level of HDL Cholesterol (mg/dL)
Lipid Profile- LDL Cholesterol | Baseline, 6 and 12 weeks
  Changes in the level of LDL Cholesterol (mg/dL)
Lipid Profile- Calculated VLDL Cholesterol | Baseline, 6 and 12 weeks
  Changes in the Calculated VLDL Cholesterol (mg/dL)
Lipid Profile- Risk Ratio (LDL/HDL) | Baseline, 6 and 12 weeks
  Changes in the Risk Ratio (LDL/HDL)
Lipid Profile- Risk Ratio (Cholesterol/HDL) | Baseline, 6 and 12 weeks
  Changes in Risk Ratio (Cholesterol/HDL)

SECONDARY OUTCOMES:
Resting Energy Expenditure | Baseline, 6 and 12 weeks
  Assessment of the Resting Energy Expenditure (REE) (kcal/day)
Resting Hemodynamics- blood pressure | Baseline, 6 and 12 weeks
  Blood pressure will be assessed before the exercise test (mmHg)
Resting Hemodynamics-Weight | Baseline, 6 and 12 weeks
  Weight (kg) will be taken before the exercise test
Resting hemodynamics- Height | Baseline, 6 and 12 weeks
  Height (m) will be taken before the exercise test
Resting hemodynamics- Fat loss | Baseline, 6 and 12 weeks
  Assessment of fat loss (kg)
Maximal Aerobic Capacity | Baseline, 6 and 12 weeks
  Milliliters of oxygen per kilogram of body weight per minute (mL/kg/min)
Musculoskeletal Strength | Baseline, 6 and 12 weeks
  One Repetition Maximum (1 RM) in pounds (lbs)
Musculoskeletal Endurance | Baseline, 6 and 12 weeks
  Number of Repetitions (#) at a given percentage of 1RM in pounds (lbs.)
Inflammatory Markers- High Sensitivity C Reactive Protein | Baseline, 6 and 12 weeks
  Changes in the level of High Sensitivity C Reactive Protein (hsCRP): mg/L
Inflammatory Markers- Aspartate Aminotransferase (AST) | Baseline, 6 and 12 weeks
  Changes in the level of Aspartate Aminotransferase : U/L
Inflammatory markers- Alanine Transaminase (ALT) | Baseline, 6 and 12 weeks
  Changes in the level of Alanine Transaminase (ALT): U/L
Inflammatory markers- Blood Urea Nitrogen (BUN) | Baseline, 6 and 12 weeks
  Changes in the level of Blood Urea Nitrogen (BUN)
Inflammatory markers- Creatinine | Baseline, 6 and 12 weeks
  Changes in the creatinine level (mg/dL)
Inflammatory markers- BUN/Creatine Ratio | Baseline, 6 and 12 weeks
  Changes in the BUN/Creatine Ratio (Ratio)
Complete Blood Count (CBC) | Baseline, 6 and 12 weeks
  CBC with differential will be measured using automated hematology analyzer. CBC parameters will be measured in their respective units (e.g., cells per microliter).
Metabolic Panel- Sodium | Baseline, 6 and 12 weeks
  Changes in Sodium level (MEQ/L)
Metabolic Panel- Potassium | Baseline, 6 and 12 weeks
  Changes in Potassium level (MEQ/L)
Metabolic Panel-Chloride | Baseline, 6 and 12 weeks
  Changes in Chloride level (MEQ/L)
Metabolic Panel- Carbon Dioxide | Baseline, 6 and 12 weeks
  Changes in the level of Carbon Dioxide (MEQ/L)
Metabolic Panel- Calcium | Baseline, 6 and 12 weeks
  Changes in the level of calcium (mg/dL)
Metabolic Panel-Protein | Baseline, 6 and 12 weeks
  Changes in the Total level of Protein (g/dL)
Metabolic Panel- Albumin | Baseline, 6 and 12 weeks
  Changes in the level of Albumin ( g/dL)
Metabolic Panel- Globulin | Baseline, 6 and 12 weeks
  changes in the level globulin (g/dL)
Metabolic Panel- Bilirubin | Baseline, 6 and 12 weeks
  Changes in the total level of Bilirubin (mg/dL)
Metabolic Panel- Alkaline Phosphatase | Baseline, 6 and 12 weeks
  Changes in the level of Alkaline Phosphatase U/L
Profile of Mood States (POMS) | Baseline, 6 and 12 weeks
  Scoring Range of -28 to 232. A higher score on the POMS indicated a greater degree of mood disturbance.
Quality of Life Assessment (QOL) | Baseline, 6 and 12 weeks
  To be evaluated using the The 36-Item Short Form Health Survey (SF-36). A higher score indicates a higher quality of life.
Cognitive function measures | Baseline, 6 weeks and 12 weeks
  The Changes in the cognitive function measures to be evaluated using the troop Color-Word test. A higher score on the Stroop indicated better performance and less interference on reading ability.

CONTACTS AND LOCATIONS:
Locations (1):
- Texas A&M University, College Station, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Martinez V, McAngus K, Dickerson BL, Leonard M, Chavez E, Chun J, Lewis M, Xing D, Gonzalez DE, Yoo C, Ko J, Rhodes H, Lee H, Sowinski RJ, Rasmussen CJ, Kreider RB. Effects of 12 Weeks of Chromium, Phyllanthus emblica Fruit Extract, and Shilajit Supplementation on Markers of Cardiometabolic Health, Fitness, and Weight Loss in Men and Women with Risk Factors to Metabolic Syndrome Initiating an Exercise and Diet Intervention: A Randomized Double-Blind, Placebo-Controlled Trial. Nutrients. 2025 Jun 19;17(12):2042. doi: 10.3390/nu17122042. PMID 40573153